CLINICAL TRIAL: NCT03886467
Title: Strategies to Increase Milk Consumption by Young Nepali Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Laurie Miller, MD, Professor of Pediatrics, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STRATEGIES
Record Dates: First submitted 2019-03-13; First posted 2019-03-22 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Child Malnutrition
Keywords: Nepal; ASF consumption
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Household clusters (separated geographically) will be randomly assigned to receive either nutrition education or to control status (no education).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education (Active Comparator): Households will participate in community-based nutrition education program specifically targeting child nutrition and milk consumption, in addition to general community development activities
  Interventions: Other: Community-based nutrition education
- Control (No Intervention): community development activities only.

INTERVENTIONS:
Other: Community-based nutrition education — Nutrition education will be included in community development training. The nutrition education will target child nutrition, particularly consumption of animal-source foods and especially milk. The importance of dietary diversity will also be emphasized. Demonstrations of food preparation techniques will also be included in the training.
  Arms: Nutrition Education

SUMMARY:
Dairy animals are an important source of income, food and nutrition security at the household level. However, substandard animal husbandry practices and limited understanding of disease prevention and control may limit dairy animal productivity. Interventions to address these issues may enhance milk production, substantially improving the well-being of smallholder farmers. In addition to increasing household income, greater milk production may improve the diet quality of household members, particularly children.

Previously, the investigators implemented a program in rural Nepal promoting enhanced animal husbandry practices (GHP), focusing on mastitis control. Concurrently, the investigators found child milk intake was strongly linked to better growth and development. However, milk intake was limited and its availability was not examined. The investigators now propose to build on these prior activities and examine strategies to increase child milk consumption. The investigators plan to introduce a nutrition education program into 200 households (with young children) which previously received GHP training. A comparison group of 200 households will serve as the control. Household surveys will be conducted at baseline and endline to assess (1) household milk production and the sustainability of adoption of GHP routines, (2) the relationship of household milk production to child milk consumption, (3) household factors influencing child milk consumption (participation in nutrition education, mother's education, socioeconomic status, etc.), and (4) longitudinal child growth and development. In addition, a pilot study will determine if households can accurately record milk production and child milk intake.

The project is designed to enhance understanding of the links between milk availability and child milk consumption in rural Nepal. It aims to explore whether milk consumption is limited by availability or other factors (nutrition awareness, socioeconomic status, maternal education). Additionally, the investigators will examine if optimization of milk consumption by young children can further boost their growth and development, and whether instruction in good animal husbandry practice and mastitis control is sustainable. These findings could more appropriately and efficiently direct resources to improve child nutrition and development and household dairy practices.

DETAILED DESCRIPTION:
The study will be conducted in close collaboration with Heifer International Nepal, a well-established branch of Heifer International, an international non-government organization based in Little Rock, Arkansas. Heifer specializes in community development activities and livestock management training; as part of Heifer's activities, participating households receive 1 or more dairy animals. The proposed study will take place in 3 districts in western Nepal (Bardiya, Surkhet, and Dang) where Heifer has been active and dairy animals have been distributed. Households (n=400) will be eligible for participation if there is at least one child between the ages of 6-66 months and at least one dairy animal. Household clusters (separated geographically) will be randomly assigned to receive either nutrition education or to control status (no education). Households assigned to control status will be offered the nutrition education after completion of data collection for the proposed project (12 months later).

The participants will be one adult in each household (usually the child's mother), and any children in the household between the ages of 6-66 months.

The study design involves 3 household visits, spaced over 12 months (thus: baseline, 6 months, and endline). In addition, information about household dairy animal milk production will be collected on a monthly basis.

At the baseline and endline household visits, the mother (or other caretaker) of the target child will be asked to respond to a questionnaire. The questionnaire will be based on standardized tools developed by "Measure Demographic and Health survey (DHS)", specifically the version used in the "2016 Nepal Demographic and Health Survey" conducted by the Government of Nepal (Ministry of Health et al. 2017) (Ministry of Health and Population Nepal et al. 2012). The questionnaire will address (A) household attributes, (B) child diet, (C) child growth, and (D) child development.

(A) Household attributes: basic demographics, possessions (used to determine wealth score by standard principal components analysis), hygiene practices, animal ownership, mother's knowledge/attitudes/practices related to child nutrition.

(B) Child diet: Consumption of animal source foods (ASFs: meat, fish, offal, eggs, or dairy) in the past 24 hours by all children in the household (ages 12-60 months) will be recorded (Ruel 2003, Steyn et al. 2007), along with the frequency of intake. The quantity of milk and other dairy foods ingested will also be determined. In addition, 16 specific foods/food groups will be documented (Kennedy et al. 2013). Milk and "other dairy products" (yogurt, paneer, cheese, etc.) will be recorded separately. In addition, the number of times in the previous week that the child consumed each of the 16 individual food items will be recorded. A diet diversity score (DDS) will be constructed by aggregating the food groups into 8 categories: starchy staples (grains and white potatoes); vitamin-A rich fruits and vegetables; other fruits and vegetables; offal, meat, and fish; eggs; legumes, nuts, and seeds; milk and dairy products; oils (Swindale et al. 2006).

(C) Child growth will also be assessed by standard anthropometric techniques (see (Miller et al. 2017) for details) using Seca scales and stadiometers and paper measuring tapes (for head and mid-upper arm circumferences).

(D) Child development: relevant sections of the Multiple Indicator Cluster Survey (UNICEF 2015), a standardized questionnaire developed by UNICEF (and validated in Nepal (Government of Nepal 2014)) to assess early child development, will be administered by the enumerator. The child's parent (usually the mother), will respond to questions related to child literacy/numeracy, gross and fine motor skills, social-emotional development, and learning skills. In addition, the age-appropriate version of the Ages and Stages Questionnaire will be administered. This simple assessment serves as a screen test for developmental issues by asking the child (or if the child is unable or unwilling to participate) to engage in developmentally appropriate activities such as completing a puzzle, jumping, scribbling with a crayon, or answering simple questions ("How old are you").

The midline visit will include only child anthropometry and child diet record.

ELIGIBILITY:
Inclusion Criteria:

* 6-66 months of age, parent willing to participate in research activity

Exclusion Criteria:

* unwillingness to participate in the research activity, plans to leave the area within the next 12 months, or child with physical or other special needs that prevent the ingestion of a normal diet-for-age.

Ages: 6 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 368 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in child height from baseline to midline | baseline, midline (0, 6 months)
  Height of children will be measured, and converted to z scores. The difference from baseline to midline will be assessed.
Change in child height from baseline to endline | baseline, endline (0, 12 months)
  Height of children will be measured, and converted to z scores. The difference from baseline to endline will be assessed.
Change in child weight from baseline to midline | baseline, midline (0, 6 months)
  Weight of children will be measured, and converted to z scores. The difference from baseline to midline will be assessed.
Change in child weight from baseline to endline | baseline, endline (0, 12 months)
  Weight of children will be measured, and converted to z scores. The difference from baseline to midline will be assessed.
Change in child head circumference from baseline to midline | baseline, midline (0, 6 months)
  Head circumference will be measured, and converted to z scores
Change in child head circumference from baseline to endline | baseline, endline (0, 12 months)
  Head circumference will be measured, and converted to z scores
Change in child development standardized score from baseline to endline | baseline and endline (0, 12 months)
  Developmental performance on standardized test, the Ages and Stages Questionnaire. The change in scores from baseline to endline will be assessed.

SECONDARY OUTCOMES:
Milk consumption by children | daily for up to 365 days
  Amount of milk consumed by children will be measured daily, using standardized measuring cups. The information will be recorded by their mothers. The daily consumption will be compiled into monthly total consumption for later analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shailes Neupane, M.S., Study Director — Valley Research Group
Locations (1):
- Valley Research Group, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No